CLINICAL TRIAL: NCT01826955
Title: Effect of Pneumoperitoneum on Cognitive Function and Regional Cerebral Oxygen
Brief Title: Effect of Pneumoperitoneum on Cognitive Function and Regional Cerebral Oxygen Saturation
Acronym: rSO2pneumo
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Jeong Kwak, Associate professor, Gachon University Gil Medical Center
Other Study IDs: GIRBA2712-2012
Record Dates: First submitted 2013-02-02; First posted 2013-04-09 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Pneumoperitoneum
Keywords: pneumoperitoneum, cognitive function
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Open gastrectomy: patient who undergoing open gastrectomy
- laparoscopic gastrectomy: patient who undergoing laparoscopic gastrectomy

SUMMARY:
The investigators hypothesized that the pneumoperitoneum with reverse Trendelenburg position could alter the rSO2 and early postoperative cognitive function.

DETAILED DESCRIPTION:
Laparoscopic gastrectomy requires a reverse-Trendelenburg position and prolonged pneumoperitoneum and it could cause significant changes in cerebral homeostasis and lead to cognitive dysfunction. We compared changes in haemodynamic variables, regional cerebral oxygen saturation, and early postoperative cognitive function in patients undergoing laparoscopic gastrectomy in the reverse Trendelenburg position with those patients that underwent conventional open gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I or II, aged 20 to 70 yrs

Exclusion Criteria:

* Patients with morbid obesity (body mass index > 30 kg/m2) or a history of cerebrovascular or respiratory disease were excluded.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who undergoing laparosopic or open gastrectomy patients who have respiratory and cardiovascular disorders were excluded
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
MMSE | 5days after end of surgery
  5 days after operation MMSE (mini-mental status exam)was recorded

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Jeong Kwak, M.D., Study Director — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

REFERENCES:
- [Background] Choi SH, Lee SJ, Jung YS, Shin YS, Jun DB, Hwang KH, Liu J, Kim KJ. Nitroglycerin- and nicardipine-induced hypotension does not affect cerebral oxygen saturation and postoperative cognitive function in patients undergoing orthognathic surgery. J Oral Maxillofac Surg. 2008 Oct;66(10):2104-9. doi: 10.1016/j.joms.2008.06.041. PMID 18848109